CLINICAL TRIAL: NCT06887023
Title: Clinicopathologic Characteristics, Progression, and Prognostic Analysis of Intraductal Papillary Neoplasm of Bile Duct
Brief Title: Clinicopathologic Characteristics, Progression, and Prognostic Analysis of IPNB
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Meng Wang, Doctor, The First Hospital of Jilin University
Other Study IDs: 2024-1244
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-02

CONDITIONS: Bile Duct Neoplasms Malignant
Keywords: intraductal papilloma of bile duct; malignancy; progression; risk factors; prognosis
MeSH Terms: conditions — Neoplasms; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main aim of this observational study is to understand the clinicopathological and prognostic information of IPNB, a rare tumor. The participants have already received treatment during their previous routine medical management and took part in follow - up. We will look into their survival information after previous medical visits and treatment.

ELIGIBILITY:
Inclusion Criteria:

* IPNB with or without malignant transformation was confirmed by pathological examination

Exclusion Criteria:

* missing other essential clinical data
* coexisting malignant tumors of other digestive system organs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients diagnosed with IPNB from eight Chinese hospitals over a 10-year period
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
death | From January 2014 to June 2024
  Died of various causes after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Jilin University, Changchun, Jililn, China